CLINICAL TRIAL: NCT05655871
Title: Investigation of the Effect of Nurse-led Transtheoretical Model-Based Video Exercise Trainings on Fall Risk to Elderly People Living in a Nursing Home
Brief Title: The Effect of Nurse-led Transtheoretical Model-Based Video Exercise Trainings on Fall Risk to Elderly People Living in Nursing Homes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Ayse Ozdemir, lecturer, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KU-AÖ-01
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Risk of Falling in the Elderly
Keywords: Nursing home; Risk of falling; Elderly individuals

STUDY DESIGN:
Intervention Model Description: There are two groups in the study, these are control and intervention groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: When creating groups in the study, the participants learned which group they belonged to, and blinding was done when the data was sent to the statistician for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enterprise Group (Experimental): Elderly individuals were divided into 5 groups according to the stages of change in the TTM scale. According to the change phase, those in the non-thinking phase are at 10:00 on Mondays, Wednesdays and Fridays, those in the thinking phase are at 13:00 on Mondays, Wednesdays and Fridays, and those in the preparatory phase are at 15:00 on Mondays, Wednesdays and Fridays of the week. They were asked to come to the seminar hall at 00:00. It was explained that a training video about physical activity would be watched. Those in the preparation phase were asked to come to the activity hall at 10:00 on Tuesdays, Thursdays and Saturdays of the week, and at 14:00 on Tuesdays, Thursdays and Saturdays of the week, while wearing their comfortable clothes. It was said that a training and motivational video about physical activity would be watched and the exercises would be done under the supervision of the researcher with the "show-and-make technique".
  Interventions: Other: Transtheoretic Model Based Video Exercise Training
- Control Group (Experimental): Data collection forms were applied to the control group in the pre-test. These forms are; "Personal Information Form, Tinetti Balance and Gait Test, Exercise Change Stages Scale, Exercise Change Process Scale, Exercise Decision-Making Scale, Exercise Self-Efficacy Scale". In order to avoid an ethical dilemma between the individuals in the control and intervention groups, the videos will be watched by the individuals in the control group at the end of the study.
  Interventions: Other: Standard Maintenance Practice

INTERVENTIONS:
Other: Transtheoretic Model Based Video Exercise Training — Initial follow-up 1-3. Between weeks 4-6, the second follow-up. Between weeks 7-9, the third follow-up. was done within weeks. Participants 10-12. No application will be made between weeks and the last test will be done in the 12th week.
  Arms: Enterprise Group
Other: Standard Maintenance Practice — Initial follow-up 1-3. Between weeks 4-6, the second follow-up. Between weeks 7-9, the third follow-up. was done within weeks. The final test will be done at week 12.
  Arms: Control Group

SUMMARY:
The aim of this study is to examine the effect of video exercise trainings based on transtheoretic model given to elderly individuals living in nursing homes under the leadership of nurses on the risk of falling in elderly individuals within nursing care programs.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of video exercise trainings based on transtheoretic model given to elderly individuals living in nursing homes under the leadership of nurses on the risk of falling in elderly individuals within nursing care programs.

This study was designed as a randomized controlled experiment. The population of the research consists of individuals aged 65 and over living in Tosya Nursing Home Elderly Care and Rehabilitation Center.

Sample size was calculated using the "G.Power-3.1.9.2" program at a 95% confidence level. As a result of the analysis, α=0.05, standardized effect size was taken from Cohen for the analysis of variance in repeated measurements with factor, due to the lack of a previous study, with a theoretical power of 0.25 to 0.95, the minimum sample size was 36 people in total, 18 control subjects. It was calculated as 18 intervention groups. However, considering that there may be data losses in the study, it was planned to recruit a total of 44 people, 22 of whom were in the control group and 22 in the intervention group, who met the inclusion criteria.

Inclusion criteria in the study

* Individuals aged 65 and over who volunteered to participate in the research
* Those with a Mini Mental Test (MMT) score ≥24
* Those with a KATZ daily living activities scale score of 6
* Does not have a cognitive/affective problem that may hinder communication Exclusion criteria from the study
* Those who have a chronic disease and cannot control it with medication (Individuals will be followed in their files.) Exclusion criteria
* The individual's desire to leave the research
* The individual has a condition that requires hospitalization
* The individual does not participate in video exercise trainings three times a week in a row.
* Death of the individual Simple randomization method was used while forming intervention and control groups in our study. In this randomization method, individuals who meet the inclusion criteria can be assigned to the groups completely randomly, with equal probability, and independently of the previous assignment, after participating in the study. Computer-assisted randomization method was used in simple randomization. For this method, the https://www.randomizer.org/ page was used and intervention and control groups were created.

Data in the research; "Standardized Mini Mental Test", "Modified Mini Mental Test for the Untrained", "KATZ Activities of Daily Living Scale", "Personal Information Form", "Tinetti Balance and Gait Test", "Exercise Change Stages Scale", "Exercise Change Process" Scale", "Exercise Decision-Making Scale", "Exercise Self-Efficacy Scale".

Before starting the research, all the elderly were invited to the nursing home seminar hall to give information about the research by meeting with the Nursing Home Director. The first interview was held with elderly individuals who could come to the seminar hall. In the first interview, information about the research was given and the compliance of the individuals with the inclusion criteria was evaluated. Written and verbal consents were obtained from the elderly individuals who met the inclusion criteria and agreed to participate in the study.

Data collection forms were applied to the intervention group in the pre-test. These forms are; "Personal Information Form, Tinetti Balance and Gait Test, Exercise Change Stages Scale, Exercise Change Process Scale, Exercise Decision-Making Scale, Exercise Self-Efficacy Scale". Elderly individuals were divided into 5 groups according to the stages of change in the TTM scale (not thinking, thinking, preparation, movement, and continuation). According to the change phase, those in the non-thinking phase are at 10:00 on Mondays, Wednesdays and Fridays, those in the thinking phase are at 13:00 on Mondays, Wednesdays and Fridays, and those in the preparatory phase are at 15:00 on Mondays, Wednesdays and Fridays of the week. They were asked to come to the seminar hall at 00:00. It was explained that a training video about physical activity would be watched. Those in the preparation phase were asked to come to the activity hall at 10:00 on Tuesdays, Thursdays and Saturdays of the week, and at 14:00 on Tuesdays, Thursdays and Saturdays of the week, while wearing their comfortable clothes. It was said that a training and motivational video about physical activity would be watched and the exercises would be done under the supervision of the researcher with the "show-and-make technique". Initial follow-up 1-3. Between weeks 4-6, the second follow-up. Between weeks 7-9, the third follow-up. was done within weeks. Participants 10-12. No application will be made between weeks and the last test will be done in the 12th week.

Data collection forms were applied to the control group in the pre-test. These forms are; "Personal Information Form, Tinetti Balance and Gait Test, Exercise Change Stages Scale, Exercise Change Process Scale, Exercise Decision-Making Scale, Exercise Self-Efficacy Scale". Initial follow-up 1-3. Between weeks 4-6, the second follow-up. Between weeks 7-9, the third follow-up. was done within weeks. The final test will be done at week 12. In order to avoid an ethical dilemma between the individuals in the control and intervention groups, the videos will be watched by the individuals in the control group at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over who volunteered to participate in the research
* Those with a Mini Mental Test (MMT) score ≥24
* Those with a KATZ daily living activities scale score of 6
* Does not have a cognitive/affective problem that may hinder communication

Exclusion criteria from the study

* Those who have a chronic disease and cannot control it with medication (Individuals will be followed in their files.) Exclusion criteria
* The individual's desire to leave the research
* The individual has a condition that requires hospitalization
* The individual does not participate in video exercise trainings three times a week in a row.
* Death of the individual

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-16 (Estimated); Study Completion 2023-01-06 (Estimated)

PRIMARY OUTCOMES:
Tinetti Balance and Gait Test | Three weeks
  Three values are given in the scoring of the Tinetti Balance and Gait Test, 0 -1-2. 0 points represents the maximum impairment (not being able to perform the movement), 1 point represents the adaptation of the specified movement, 2 points independence (the movement is done as desired). Individual scores are then combined to form three measures, the overall gait assessment score, the overall balance assessment score, and the sum of the gait and balance scores. The maximum score that can be obtained for the walking assessment is 12. The maximum score that can be obtained for the balance assessment is 16. The maximum total score that can be obtained from the Tinetti Balance and Gait Test is 28. In general, a total score of ≤18 indicates a high risk of falling, a range of 19-24 indicates a medium fall risk and a score of ≥24 indicates a low risk of falling.
Exercise Stages of Change Scale | Three weeks
  It consists of 5 stages: not thinking, thinking, preparing, acting and continuing.

SECONDARY OUTCOMES:
Exercise Change Process Scale | 1st week, 9th week and 12th week
  The scale of the change process; It is a 40-item scale consisting of 10 sub-dimensions, five of which are cognitive processes and five are behavioral processes. The five-point Likert scale evaluates the previous month. The items of the scale range from one to five points. While the highest score that can be obtained from the scale is 200, the lowest score is 40. An increase in the scale score indicates that individuals progress positively in the exercise change process.
Exercise Decision Making Scale | 1st week, 9th week and 12th week
  The scale, which consists of 16 questions, is a five-point Likert type. The first 10 questions measure the perception of benefit, while the last six questions measure the perception of harm. While the lowest score that can be taken from the perception of benefit sub-dimension of the decision-making scale is 10 and the highest score is 50, the lowest score that can be obtained from the perception of harm sub-dimension is 6 and the highest score is 30. In order for the individual to be successful in change, it is expected that the benefit perception score will increase and the harm perception score will decrease.
Exercise Self-Efficacy Scale | 1st week, 9th week and 12th week
  Exercise self-efficacy scale is five-item and five-point Likert type. The highest score that can be obtained from the scale is 25, and the lowest score is 5. The increase in the scale score indicates that the individuals' self-efficacy for exercising has improved.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Özdemir, Instructor, Principal Investigator — PhD Thesis Student; Ayla Demirtaş, Associate professor, Study Director — PhD Thesis Advisor
Locations (1):
- Kastamonu University, Kastamonu, Tosya, Turkey (Türkiye)